CLINICAL TRIAL: NCT07161687
Title: HYMPAVZI S.C. INJECTION 150 mg Pen SPECIAL INVESTIGATION
Brief Title: A Study to Learn About the Study Medicine -Hympavzi in Congenital Hemophilia Patients Without Inhibitors in Japan.
Acronym: HIZ
Status: Active, not recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B7841012
Record Dates: First submitted 2025-09-02; First posted 2025-09-09 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Hemophilia A or B
Keywords: Marstacimab,Hympavzi,Hemophilia
MeSH Terms: conditions — Hemophilia A | interventions — marstacimab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Marstacimab: hemophilia patients without inhibitor
  Interventions: Drug: Marstacimab

INTERVENTIONS:
Drug: Marstacimab — For patients aged 12 years or older and weighing at least 35 kg, marstacimab is administered subcutaneously at a dose of 300 mg as the initial dose, followed by 150 mg once weekly. If the patient weighs 50 kg or more and shows an inadequate response, the dose may be increased to 300 mg once weekly for subcutaneous administration.
  Other Names: Hympavzi

SUMMARY:
A study to evaluate the safety of Hympavzi under the actual use in patients with congenital hemophilia who do not have inhibitors.

DETAILED DESCRIPTION:
The objective of this study is to assess the safety of this drug under actual usage conditions in patients with congenital hemophilia who do not have inhibitors.

The observation period will be up to three years. However, for cases in which administration of the drug is discontinued, information will be collected up to the point of discontinuation.

ELIGIBILITY:
Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

* Patients who have received at least one dose of this drug after the launch of this drug

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who have received at least one dose of this drug after the launch of this drug.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2025-10-30 (Actual); Primary Completion 2029-12-13 (Estimated); Study Completion 2029-12-13 (Estimated)

PRIMARY OUTCOMES:
Number of the participants with adverse drug reactions | The evaluation period is from the first dose of Himpavzi up to 156 weeks (3 years).
  An adverse drug reaction (ADR) was a treatment-related adverse event, and any untoward medical occurrence attributed to Himpavzi in a participant who received Himpavzi. A serious adverse drug reaction (SADR) was a treatment-related adverse event resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening; initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect. Relatedness to Himpavzi was assessed by the physician.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Inc, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7841012